CLINICAL TRIAL: NCT01135680
Title: Double-Blind Randomized Placebo-Control Trial to Evaluate Electrocardiogram Effects of HPN-100 as Defined by Clinical and Supratherapeutic Dose in Healthy Men and Women
Brief Title: Double-Blind Randomized Crossover Trial to Access Electrocardiogram Effects of HPN-100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HPN-100-010
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Drug Toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — glycerol phenylbutyrate; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Placebo Comparator): Cohort A: 9 mL HPN-100 or placebo
  Cohort B: 12 mL HPN-100 placebo
  Interventions: Drug: HPN-100; Drug: HPN-100 or Placebo
- Arm 2 (Placebo Comparator): This study requires 4 periods. In each of the periods you will receive one of the dose groups listed below. At the completion of the study you will have participated in all 4 dose groups. The order in which you participate in each dose group will be randomly assigned.
  Dose Group A: 9 mL placebo via oral syringe 3 times daily for 3 days
  Dose Group B: single oral dose of 400 mg moxifloxacin on study Day 3
  Dose Group C: 6 mL HPN-100 and 3 mL placebo via oral syringe 3 times daily for 3 days
  Dose Group D: 9 mL HPN-100 via oral syringe 3 times daily for 3 days
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: HPN-100

INTERVENTIONS:
Drug: HPN-100 — single oral dose of 9 mL HPN-100 given via syringes 3 times daily for 3 days
  Arms: Arm 1
Drug: HPN-100 or Placebo — single oral dose of 12 mL HPN-100 given via syringes 3 times daily for 3 days
  Arms: Arm 1
Drug: Placebo — single oral (by mouth) dose of 9 mL placebo given via syringes 3 times daily for 3 days
  Arms: Arm 2
Drug: Moxifloxacin — single oral 400-mg dose on study Day 3
  Arms: Arm 2
Drug: HPN-100 — single oral dose of 6 mL HPN-100 and 3 mL placebo given via syringes 3 times daily for 3 days
  Arms: Arm 2
Drug: HPN-100 — single oral dose of 9 mL HPN-100 given via syringes 3 times daily for 3 days
  Arms: Arm 2

SUMMARY:
Arm 1:

Primary Objective:

• To determine the safety and tolerability of multiple ascending, supratherapeutic doses of HPN-100.

Arm 2:

Primary Objective:

• To assess the effects of steady-state levels of HPN-100 metabolites (4 phenylbutyric acid [PBA], phenylacetic acid [PAA], and phenylacetylglutamine [PAGN]) on 12-lead electrocardiogram (ECG) parameters in healthy male and female subjects with the primary endpoint being the time-matched change from baseline in the QT interval corrected for heart rate (HR) based on an individual correction method (QTcI).

DETAILED DESCRIPTION:
Assess the effects of steady-state levels of HPN-100 metabolites (4-phenylbutryic acid (PBA), phenylacetic acid (PAA), and phenylacetylglutamine (PAGN) on 12-lead electrocardiogram (ECG) parameters in health male and female subjects with the primary endpoint being the time-matched change from baseline in the QT interval corrected for heart rate(HR) based on an individual correction method (QTcl).

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good health
* Negative hepatitis panel and negative HIV antibody screens
* Females must be non-pregnant, non-lactating, and either postmenopausal or agree to to use adequate contraceptive methods throughout the study
* Males must either be sterile or willing to use adequate contraceptive methods throughout the study
* Willing and able to comply with all trial requirements
* Able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

* History or clinical manifestations of significant allergic, metabolic, hepatic, renal, endocrine, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders
* History of hypersensitivity or allergies to any drug compound
* History of stomach or intestinal surgery or resection
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction within 1 year
* Use of any tobacco-containing or nicotine-containing products within 3 months
* Participated in any other clinical trial of an investigational drug (or a medical device) within 30 days
* Use of any prescription medications/products other than contraceptives within 14 days
* Use of any over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days
* Test positive for drug(s) of abuse, ethanol, or cotinine
* Have donated blood or blood components within 30 days
* Have received blood products within 2 months
* Have a history of unexplained syncope
* Have a family history of unexplained sudden death

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the rate and severity of adverse events in each treatment group. | 3-day treatment period
Changes from baseline QTcI as a measure of effects of study-state HPN-100 metabolites: PBA, PAA, and PAGN | 4 treatment regimens for 3 days with a 4 day minimum washout period between treatments

SECONDARY OUTCOMES:
Correlate time-matched ECG waveform changes to steady-state levels of HPN-100 by using QTcB and QTcF formulas to assess ECG morphologic changes. | 4 treatment regimens for 3 days with a 4 day minimum washout period between treatments
Correlate time-matched QTcI change from baseline and serum levels of PBA, PAA, and PAGN drawn on Day 1, Day 2, Day 3, and Day 4 | 4 treatment regimens for 3 days with a 4 day minimum washout period between treatments
Gender differences in metabolism of HPN-100 as measured by time-matched serum levels of HTN-100, PBA, PAA, and PAGN via samples drawn on Day 1, Day 2, Day 3, and Day 4. | 4 treatment regimens for 3 days with a 4 day minimum washout period between treatments
Number and severity of adverse events in each treatment group. | 4 treatment regimens for 3 days with a 4 day minimum washout period between treatments

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Pharmacology, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing